CLINICAL TRIAL: NCT06347055
Title: Neuronavigated Non-invasive Brain Stimulation for Nicotine Dependence.
Brief Title: NeuroControl of Nicotine Dependence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Froeliger, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 403690
Record Dates: First submitted 2024-03-20; First posted 2024-04-04 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Nicotine Dependence
Keywords: Tobacco; Smoking; TMS; fMRI; Nicotine; Cognitive Control
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- cTBS to Ventrolateral Prefrontal Cortex (Experimental): Continuous theta-burst stimulation (cTBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. cTBS will be applied to the ventrolateral prefrontal cortex.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- cTBS to Dorsomedial Prefrontal Cortex (Experimental): Continuous theta-burst stimulation (cTBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. cTBS will be applied to the dorsomedial prefrontal cortex.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- cTBS to Vertex (Experimental): Continuous theta-burst stimulation (cTBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. cTBS will be applied to the vertex.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Continuous theta burst rTMS
  Other Names: cTBS

SUMMARY:
The purpose of the study is to examine the effects of continuous theta burst stimulation (cTBS) on different forms of cognitive control in adults who smoke cigarettes, and to determine if the location where cTBS is delivered may help smokers reduce or quit smoking. Participation in the study will take 3-weeks over 4 visits, with a total time commitment of approximately 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Nicotine Dependence as measured by: Smoke ≥ 8 cigarettes/day for ≥ 2 yrs, expired carbon monoxide (CO) concentration of ≥ 10 ppm, positive urine cotinine test and FTND score ≥ 3 Or ≥ 15 uses of electronic cigarette/day for ≥ 1 year, positive urine cotinine test, and PS-ECDI score ≥ 3
2. English Fluency
3. Functional Vision (with corrective lenses as needed)

Exclusion Criteria:

1. Use of psychotropic and antiepileptic medications in the last month
2. Presence of an untreated illness or serious medical condition
3. History of major neurological illness
4. Contraindication to TMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for >15 min., implanted electronic device, metal in the head) or MRI.
5. Any use of substances that lower seizure threshold.
6. Current or past psychosis
7. Electroconvulsive therapy in the past 6 months
8. Unstable cardiac disease or hypertension, severe renal or liver insufficiency, or sleep apnea
9. BAC greater than 0.0.
10. Positive urine pregnancy test
11. Any other concern that in the investigator's opinion would impact participant safety, study instruction compliance, or confound the interpretation of the study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-03-25 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Acute effects of cTBS on cognitive control | 1 hour after receiving cTBS
  between-arm differences in neurocognitive task performance as measured by percent correct on an inhibitory control task and self reported craving on a regulation of craving task.

SECONDARY OUTCOMES:
Exploratory: Acute effects of cTBS on fMRI brain response | 1 hour after receiving cTBS
  between-arm differences in whole brain fMRI BOLD functional connectivity. Neural network connectivity will be characterized using rZ values.

OTHER OUTCOMES:
Safety and Tolerability | 24 hours following receipt of cTBS
  Safety and tolerability of cTBS administered to each cortical location, as measured by self reported side effects on a review of symptoms questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Neuroscience Center, Columbia, Missouri, United States